CLINICAL TRIAL: NCT03721809
Title: Characterization of the Inflammatory Profile of Patients With Macrophage Activation Syndrome Secondary to Bacterial Sepsis
Acronym: SAMOKINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017/185/HP
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Macrophage Activation Syndrome
MeSH Terms: conditions — Macrophage Activation Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- macrophage activation syndrome secondary to bacterial sepsis (Other): Patients hospitalized in medical intensive care for macrophage activation syndrome secondary to bacterial sepsis
  Interventions: Biological: Blood samples
- bacterial sepsis/septic shock (Other): Patients hospitalized in medical intensive care for sepsis / septic shock
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — There are 3 specific blood sampling times for each patient, on D1, D2 and D5 (D1 being the day of inclusion): cytokine samples (IL-1β, IL-6, IL-10, TNF-α, IFN-gamma) on 5ml dry tube.
  On D1, a 2.5ml PAXgene tube will also be taken for each patient.

SUMMARY:
The pathophysiology of macrophage activation syndrome has been mainly studied in pediatric genetic primary forms. There is little data in secondary forms related to bacterial sepsis. Because of the seriousness of this entity (43% of deaths in intensive care in the largest cohort published so far by the medical resuscitation team of Rouen University Hospital), it is necessary to better understand the physiopathological mechanisms to be able to propose a suitable therapy. For now, the management of this syndrome is far from consensual. Some authors advocate a single etiological treatment, while others suggest the need for intensive management of anti-inflammatory and immunosuppressive type. The fragility of resuscitation patients does not allow intensive immunosuppressive therapies as proposed by some authors. In the era of immunotherapy, the precise knowledge of physiopathological data would make it possible to propose a targeted therapy with little risk of adverse effects. Recent work has indeed shown excellent tolerance of immunotherapy during sepsis and could be applied eventually in patients with macrophage activation syndrome.

ELIGIBILITY:
Inclusion Criteria:

Patient hospitalized in intensive care for macrophage activation syndrome secondary to sepsis / bacterial septic shock with a strong clinical probability score (defined by a HScore> 80% cf appendix 4) (experimental population) or Patient hospitalized in intensive care for sepsis or septic shock (control population)

* Age ≥ 18 years
* Person affiliated with a social security scheme or beneficiary of such a scheme
* Trusted person or informed patient who has signed the consent to participate in the research. (If the patient is unable to sign his / her consent (emergencies) the consent will be signed by the person of trust, and consent to further study will be requested from the patient).
* Effective contraception in women of childbearing potential (negative pregnancy test). For postmenopausal women, a confirmation diagnosis should be obtained (amenorrhea for at least 12 months before the inclusion visit).

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Person deprived of liberty by an administrative or judicial decision
* Protected major subject, under tutorship or curatorship
* Patient participating in another interventional clinical trial with the same primary objective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
quantitative measurement of plasma IL-1β in MAS patients secondary to septic sepsis / bacterial septic shock in comparison with a control population of sepsis /septic shock. | performed on day 1
  measured by the luminex method

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rouen, Rouen, France